CLINICAL TRIAL: NCT06239246
Title: Analyzing the Association Between Cardiovascular Diseases and Mental Illness Considering Environmental Risk Factors
Brief Title: Association Between Cardiovascular Diseases and Mental Illness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-R062
Record Dates: First submitted 2023-12-25; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Cardiovascular Diseases; Mental Disorder
MeSH Terms: conditions — Cardiovascular Diseases; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 2000 hospitalized patients: hospitalized patients with heart diseases
  Interventions: Other: Behavioral
- 10000 community population

INTERVENTIONS:
Other: Behavioral — Psychotherapy: Cognitive-behavioral therapy (CBT), Internet-based cognitive-behavioral therapy (I-CBT), cognitive-behavioral therapy for insomnia (CBT-I), self-management education for heart failure, "blended" intervention; Drug treatment (cardiovascular drugs: aspirin, clopidogrel, ticagrelor, statins; psychiatric drugs: SSRIs, SNRIs, etc.);
  Groups: 2000 hospitalized patients

SUMMARY:
Cardiovascular diseases (CVD) are important public health concerns around the world and closely associated with the development and progression of mental illness, which in turn increases the risk of developing cardiovascular diseases. This study aimed (1) to explore the known or unknown protective and risk factors underlying this comorbidity using questionnaires; (2) to study the biomarkers (body fluid, imaging) of the participants, and to find the influence on the relationship between CVD and mental health; (3) to identify high-risk populations for mental disorders in CVD patients and to establish prediction models. (4) to establish a specialized medical database.

DETAILED DESCRIPTION:
Patients with depression and cardiovascular comorbidities have a worse prognosis, a sharply reduced quality of life, and a much higher incidence of fatal CVD events, such as acute infarction, than patients with a single disease. However, due to the variety of potential causative factors and clinical manifestations, population variability, long duration of the disease, as well as neurological disorders of the exact causative mechanism still unclear, the psychological assessment among patients with cardiovascular diseases is remarkably inadequate studied.

In this study, two cohorts are established that include 2000 hospitalized patients and 5000 of the entire population. All individuals are screened for depression and anxiety. Those who score positive will be advised to enroll in this study. Patients are then randomized to receive collaborative care involving the patient, the patient's primary care physician, cardiologist and nurse case manager, or usual care is defined for each patient. Whole blood and serum samples are obtained from all patients, which will be measured for a panel of metabolic and inflammatory indicators. Patients in both cohorts will be monitored for depression severity and duration at 6 and 12 months after enrollment. A statistical technique is applied to determine the effect size of potential risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient and inpatient cardiology patients, diagnosed with at least one cardiovascular disease and at least one psychological disorder
2. Cardiovascular diseases: ACS (STEMI, non-STEMI, unstable angina), arrhythmia (atrial fibrillation, atrioventricular block), heart failure (stable/unstable), hypertension, cardiomyopathy (hypertrophic, dilated)
3. Psychological disorders: structured interview diagnosed as depression, anxiety, insomnia; PHQ-9/GAD-7 score ≥ 10 points.

4．18-70 years old

Exclusion Criteria:

1. Clear suicidal ideation: PHQ-9 item 9 suicide ideation ≥ 3 points
2. Severe mental illnesses such as bipolar disorder, schizophrenia
3. Currently under psychotherapy
4. Severe cardiovascular diseases or other severe chronic life-threatening diseases
5. Refusal to participate
6. Abuse of alcoholism and drugs
7. Pregnant or breastfeeding
8. Cognitive impairment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals aged 18 to 75 years old who had normal cognition.
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
severity of depressive symptoms through CES-D | cross-sectional analyses in 2024
  severity of depressive symptoms through CES-D Include 20 questions, sum all points. Total points 60. Judgment critaria: ≤15 as no depressive symptoms, 16-19 as possible depressive symptoms, ≥20 as definite depressive symptoms.
The Patient Health Questionnaire 9-item depression scale (PHQ-9) | cross-sectional analyses in 2024
  Total points 27. depression judgment criteria: 0-4 as no, 5-9 as mild, 10-14 as moderate, 15-19 as moderate to severe, 20-27 as severe.
  Framingham risk score,NYHA cardiac function classification, six-minute walk test
7-item Generalized Anxiety Disorder scale (GAD-7) | cross-sectional analyses in 2024
  Total points 21. Anxiety judgment criteria: 0-4 as no, 5-9 as mild, 10-14 as moderate, 15-21 as severe.
Pittsburgh sleep quality index,PSQI | cross-sectional analyses in 2024
  Include 23 items. Total points 21. Sleep quality judgment criteria: 0-5 very good, 6-10 good, 11-15 fair, 16-21 poor.
New York heart failure classification | cross-sectional analyses in 2024
  Judgment criteria:
  Class I: patients are not limited in daily activities; Class II: patients are mildly limited in physical activity; Class III: patients are significantly limited in physical activity; Class IV: patients can not be engaged in any physical activity.
Six-minute walk test | cross-sectional analyses in 2024
  A 6-minute walking distance of less than 150 meters indicates severe heart failure, 150-450 meters indicates moderate heart failure, and>450 meters indicates mild heart failure.

SECONDARY OUTCOMES:
Major Adverse Cardiac Events | 24 months
  Hospitalization or mortality from Major Adverse Cardiac Events

CONTACTS AND LOCATIONS:
Overall Officials: Ruan Liemin, Study Director — Department of Psychosomatic Medicine
Locations (1):
- the first affliliated hospital of Ningbo University, Ningbo, Zhejiang Province, China, Ningbo, Zhejiang, China

REFERENCES:
- [Derived] Wu Y, Mi Y, Cui H, Song Q, Ruan L. Relationship between recurrently elevated hsCRP and adverse cardiovascular events among depressed patients in China: a time-to-event analysis. Front Cardiovasc Med. 2025 Oct 17;12:1554897. doi: 10.3389/fcvm.2025.1554897. eCollection 2025. PMID 41179571